CLINICAL TRIAL: NCT07380958
Title: Mirror Therapy as an Adjunct to Rehabilitation Following Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Marissa Hanlon, Assistant Professor, Department of Physical Therapy Education, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2384397-1
Record Dates: First submitted 2026-01-09; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Total Knee Arthroplasty Recovery
Keywords: Total knee replacement; pain; mirror therapy; range of motion; joint replacement; rehabilitation following a knee replacement
MeSH Terms: conditions — Pain | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham, no mirror provided (Sham Comparator): Subjects will participate in ROM activities, consistent with standard PT care, without a mirror
  Interventions: Other: Sham Intervention
- Active mirror (Experimental): Subjects will participate in ROM activities, consistent with standard PT care, with a mirror
  Interventions: Other: Mirror Therapy

INTERVENTIONS:
Other: Mirror Therapy — Using a mirror while participating in ROM activities.
  Arms: Active mirror
Other: Sham Intervention — Using a covered mirror, unable to see reflection. subject will perform all ROM activities
  Arms: Sham, no mirror provided

SUMMARY:
The investigators are looking to see if using a mirror during knee exercises after a knee replacement helps participants with less pain and/or better knee range of motion.

DETAILED DESCRIPTION:
Purpose: To examine the effectiveness of mirror therapy combined with standard care physical therapy on knee range of motion (ROM), pain levels, and physical function in individuals following a total knee arthroplasty (TKA).

Background: Following a TKA, patients often present with numerous impairments including joint stiffness, pain, decreased strength, and impaired mobility. These limitations can inhibit functional progress during rehabilitation and recovery. Mirror therapy is a potential treatment option that may assist in reducing these impairments and improving recovery following TKA.

Study Activities: Active and sham group activities will add-on to the physical therapy session and are considered part of standard care, with no change to the current billing process. Both groups will participate in ROM activities, consistent with standard PT care, as part of a billable treatment. The active group with do standard practice ROM activities while looking at a mirror and the sham group will perform ROM activities without a mirror.

Interventions:

* Treatment will start within 2 weeks (14 days) of the total knee replacement.
* There will be 8 sessions within a 4-week time frame.

Data Analysis: Demographic information will be reported using descriptive statistics. Analyses will use linear mixed-effects models with fixed effects for Group, Time, and the Group × Time interaction, and with subject-level random effects to account for repeated measures. The primary inference will be the Group × Time interaction.

ELIGIBILITY:
Inclusion Criteria:

1. Candidates that have been screened and deemed eligible for a TKA and received a TKA 14 days or less post operation.
2. English speaking
3. Able to understand and follow instructions
4. Has at least 5 degrees of knee extension to 100 degrees of knee flexion AROM on the contralateral knee
5. Able to perform unilateral stance on contralateral side for at least 5 seconds (balance assistance allowed)
6. Able to perform exercises

Exclusion Criteria:

1. Post-surgical complications (DVT, infection, nerve injury, vascular injury)
2. Pain rating on NPRS no more than a 4/10 on the contralateral LE
3. Significant scar or deformity of the contralateral LE
4. Visual impairments causing an inability to see the reflection in a mirror

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Pain NRS (Pain Numerical Rating Scale) | Every visit, visits 1, 2, 3, 4, 5, 6, 7 & 8. Visits start within 14 days of the TKA and occur a total of 8 times within a 4 weeks time frame.
  Subject rates pain from 0-10 with 0 being no pain and 10 being the worst pain
Knee Flexion and Extension Goniometry | Every visit, visits 1, 2, 3, 4, 5, 6, 7 & 8. Visits start within 14 days of the TKA and occur a total of 8 times within a 4 weeks time frame.
  A measurement of knee flexion and knee extension, using a goniometer, will be completed.

SECONDARY OUTCOMES:
Gait Speed | Visit 1 and visit 8. Visits start within 14 days of the TKA and occur a total of 8 times within a 4 weeks time frame.
  Subject's gait speed will be measured in meters/second.
Knee Injury and Osteoarthritis Outcome Score, Junior (KOOS Jr) | Visit 1 and visit 8. Visits start within 14 days of the TKA and occur a total of 8 times within a 4 weeks time frame.
  Knee Injury and Osteoarthritis Outcome Score, Junior (KOOS Jr) is a short, 7-question survey used by doctors to quickly assess a patient's knee pain, stiffness, and daily function. The raw score is converted to a 0-100 scale with a score of 0 = total disability and 100 = full function without pain.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toshmniwal, P., Wani, Dr. S., Mungikar, Dr. S., Garg, Dr. K., & Katage, Dr. G. (n.d.). Effectiveness of mirror therapy in adjunct to conventional physiotherapy on pain, instability, joint mobility, and proprioception in patients with post anterior cruciate ligament reconstruction surgery: a randomized controlled trial. Neuro Quantology, 20(9), 5954-5960.
- [Background] Ramachandran, V. S., et al. "Touching the Phantom Limb." Nature, vol. 377, no. 6549, Oct. 1995, pp. 489-490, https://doi.org/10.1038/377489a0
- [Background] Frenkel MO, Maltese S, Mayer J, Thermann H. Does mental practice supplemented by mirror therapy promote flexion ability after total knee endoprosthesis? Physical Medicine and Rehabilitation Research. 2018;3(2):1-10.
- [Background] Ray L. Joint Replacement Surgery. rheumatology.org. Published February 2024. https://rheumatology.org/participants/joint-replacement-surgery
- [Background] Rebne E, Louw A, Podalak J, et al. Mirror Therapy for Total Knee Arthroplasty: A Pilot Study. Surgery Research Journal. 3(1):1-9.
- [Background] Nishi K, Moriuchi T, Okamura R, Hasegawa T, Chang X, Matsumoto S, Koseki H, Higashi T. Mirror Therapy Reduces Pain and Preserves Corticomotor Excitability in Human Experimental Skeletal Muscle Pain. Brain Sci. 2024 Feb 23;14(3):206. doi: 10.3390/brainsci14030206. PMID 38539595